CLINICAL TRIAL: NCT06619600
Title: Effect of Dapagliflozin in Myocardial Fibrosis and Ventricular Function in Patients With a ST-segment Elevation Myocardial Infarction
Acronym: DAPA-STEMI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESR-19-14489; 2018-003105-25 (EudraCT Number)
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-09

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI); Diabetes Mellitus; Heart Failure; Myocardial Fibrosis
Keywords: Dapagliflozin; Myocardial Fibrosis; ST-segment Elevation Myocardial Infarction (STEMI); Cardiac Magnetic Resonance (CMR); Heart Failure
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Diabetes Mellitus; Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg qd
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Matched placebo qd
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg qd
  Arms: Dapagliflozin
Drug: Placebo — Matched placebo qd
  Arms: Placebo

SUMMARY:
The DAPA-STEMI trial investigates whether dapagliflozin, a sodium-glucose cotransporter 2 inhibitor (SGLT2i), reduces heart muscle scarring (fibrosis) and improves heart function after a ST-segment elevation myocardial infarction (STEMI). The trial will use cardiac MRI to measure changes in heart structure and function over six months. Patients aged 30-85 who have had a recent STEMI will receive either dapagliflozin or a placebo. The study aims to provide mechanistic insights into heart failure prevention after heart attacks.

DETAILED DESCRIPTION:
The DAPA-STEMI trial is a clinical research study designed to investigate whether dapagliflozin, a medication known as a sodium-glucose cotransporter 2 inhibitor (SGLT2i), can reduce the extent of heart muscle damage and improve heart function in patients who have experienced a heart attack. Specifically, the study focuses on patients who have had a type of heart attack known as a ST-segment elevation myocardial infarction (STEMI), which is a serious condition that often leads to long-term heart damage and heart failure.

The study aims to answer whether treatment with dapagliflozin can reduce the amount of scarring (fibrosis) that develops in the heart after a heart attack, and whether this reduction in scarring improves the overall function of the heart. Scarring in the heart can lead to stiffening of the heart muscle, which affects its ability to pump blood effectively and can result in heart failure. By using advanced imaging techniques, such as cardiac magnetic resonance imaging (MRI), the study will measure changes in the heart's structure and function over time.

The primary question the study seeks to answer is whether dapagliflozin can decrease the amount of heart muscle scarring (fibrosis) and improve heart function when compared to a placebo (an inactive treatment). The study will also examine whether dapagliflozin affects other important heart health markers, such as blood levels of proteins that indicate heart muscle damage and the overall size and function of the heart chambers.

The study will enroll patients aged 30 to 85 who have recently experienced a STEMI and undergone successful treatment to open the blocked artery. Participants will be randomly assigned to receive either dapagliflozin or a placebo for six months, and their heart function and scarring will be monitored through imaging and blood tests during that time.

The results of this study may provide important insights into new ways to protect the heart after a heart attack and prevent the development of heart failure, offering potential benefits to a wide range of patients who experience heart attacks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 30 - 85 years of age.
2. Patients with first infarction with ST-segment elevation documented in an ambulance or a cardiac catheterization laboratory (ST-segment elevation ≥2 mm in at least two contiguous leads) less than 12 hours after onset of symptoms that last ≥ 20 min, that is treated with primary percutaneous cardiac intervention.
3. The target lesion must be a de novo lesion located in a native vessel.
4. The patient understands and accepts the clinical monitoring and cardiac magnetic resonance.
5. The patient has to be hemodynamically stable (Killip classification 1) at the time of the initial cardiac magnetic resonance.
6. A left ventricular ejection fraction ≤50% in the baseline echocardiogram.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Type 1 diabetes.
3. Previous treatment with SGLT2i.
4. Severe liver disease (Child-Pugh C).
5. Kidney disease defined as stage III or worse (eGFR less than 45 ml/min).
6. Systolic blood pressure less than 90 mmHg at the screening visit.
7. Malignancy (receiving active treatment) or other life-threatening diseases.
8. Any contraindication to cardiac MRI (e.g., claustrophobia, metal implants, penetrating eye injury, or exposure to metal fragments in the eye that require medical attention).
9. Previous complicated urinary tract infection in men or repeated urinary infection in women.
10. Patients treated with fibrinolytic therapy.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Extracellular volume (ECV, %) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the extracellular volume (ECV) of the remote myocardium between the 6-month and baseline follow- up, evaluated by cardiac magnetic resonance (ΔECV dapagliflozin group versus ΔECV placebo group; [ΔECV = ECV 6-month - ECV baseline]).

SECONDARY OUTCOMES:
Serum levels of C-terminal propeptide of type I procollagen (PICP) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the serum levels of C-terminal propeptide of type I procollagen (PICP) between the 6-month and baseline follow- up (ΔPICP dapagliflozin group versus ΔPICP placebo group; [ΔPICP = PICP 6-month - PICP baseline]).
N-terminal propeptide of type III (PIIINP) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the serum levels of N-terminal propeptide of type III (PIIINP) between the 6-month and baseline follow- up (ΔPIIINP dapagliflozin group versus ΔPIIINP placebo group; [ΔPIIINP = PIIINP 6-month - PIIINP baseline]).
Galectin-3 procollagen (Gal-3) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the serum levels of galectin-3 procollagen (Gal-3) between the 6-month and baseline follow- up (ΔGal-3 dapagliflozin group versus ΔGal-3 placebo group; [ΔGal-3 = Gal-3 6-month - Gal-3 baseline]).
High-Sensitivity cardiac Troponin I (hs-cTnI) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the serum levels of High-Sensitivity cardiac Troponin I (hs-cTnI) between the 6-month and baseline follow- up (hs-cTnI dapagliflozin group versus hs-cTnI placebo group; [Δhs-cTnI = hs-cTnI 6-month - hs-cTnI baseline]).

OTHER OUTCOMES:
N-terminal pro-brain natriuretic peptide (NT-proBNP) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the serum levels of N-terminal pro-brain natriuretic peptide (NT-proBNP) between the 6-month and baseline follow- up (NT-proBNP dapagliflozin group versus NT-proBNP placebo group; [ΔNT-proBNP = NT-proBNP 6-month - NT-proBNP baseline]).
Soluble suppression of tumorigenicity 2 (sST2) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the serum levels of Soluble suppression of tumorigenicity 2 (sST2) between the 6-month and baseline follow- up (sST2 dapagliflozin group versus sST2 placebo group; [ΔsST2 = sST2 6-month - sST2 baseline]).
Indexed ventricular mass of the left ventricle (LVMI, g/m^2) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the Indexed ventricular mass of the left ventricle (LVMI) between the 6-month and baseline follow- up, evaluated by cardiac magnetic resonance (ΔLVMI dapagliflozin group versus ΔLVMI placebo group; [ΔLVMI = LVMI 6-month - LVMI baseline]).
Indexed End-diastolic volume of the left ventricle (LVEDVI, mL/m^2) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the Indexed End-diastolic volume of the left ventricle (LVEDVI) between the 6-month and baseline follow- up, evaluated by cardiac magnetic resonance (ΔLVEDVI dapagliflozin group versus ΔLVEDVI placebo group; [ΔLVEDVI = LVEDVI 6-month - LVEDVI baseline]).
Indexed End-systolic volume of the left ventricle (LVESVI, mL/m^2) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the Indexed End-systolic volume of the left ventricle (LVESVI) between the 6-month and baseline follow- up, evaluated by cardiac magnetic resonance (ΔLVESVI dapagliflozin group versus ΔLVESVI placebo group; [ΔLVESVI = LVESVI 6-month - LVESVI baseline]).
Left ventricular ejection fraction (LVEF, %) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the Left ventricular ejection fraction (LVEF) between the 6-month and baseline follow- up, evaluated by cardiac magnetic resonance (ΔLVEF dapagliflozin group versus ΔLVEF placebo group; [ΔLVEF = LVEF 6-month - LVEF baseline]).
Body weight (BW, Kgs) | 6 months
  To determine the effect of dapagliflozin compared with placebo in the change (Δ) of the Body weight (BW) between the 6-month and baseline follow- up, (ΔBW dapagliflozin group versus ΔBW placebo group; [ΔBW = BW 6-month - BW baseline]).
Major Adverse Cardiovascular Events (MACE) | 6 months
  Difference in the incidence of Major Adverse Cardiovascular Events (MACE), defined as a composite of death, non-fatal myocardial infarction, and non-fatal stroke, between the dapagliflozin and placebo groups.
Hospitalizations for Heart Failure (HHF) | 6 months
  Difference in the incidence of Hospitalizations for Heart Failure (HHF) between the dapagliflozin and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Ortega, MD, PhD, Principal Investigator — Division of Cardiology, University of Florida College of Medicine-Jacksonville, Jacksonville, Florida, USA.; Salvatore Brugaletta, MD, PhD, Study Chair — Hospital Clínic, Cardiovascular Clinic Institute, Institut d'Investigacions Biomèdiques August Pi i Sunyer (IDIBAPS), University of Barcelona, Barcelona, Spain.
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Clinic of Barcelona, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: Undecided
To be discussed.

REFERENCES:
- [Background] Perea RJ, Morales-Ruiz M, Ortiz-Perez JT, Bosch X, Andreu D, Borras R, Acosta J, Penela D, Prat-Gonzalez S, de Caralt TM, Martinez M, Morales-Romero B, Lasalvia L, Donnelly J, Jimenez W, Mira A, Mont L, Berruezo A. Utility of galectin-3 in predicting post-infarct remodeling after acute myocardial infarction based on extracellular volume fraction mapping. Int J Cardiol. 2016 Nov 15;223:458-464. doi: 10.1016/j.ijcard.2016.08.070. Epub 2016 Aug 8. PMID 27544605
- [Background] Ortega-Paz L, Cristobal H, Ortiz-Perez JT, Garcia de Frutos P, Mendieta G, Sandoval E, Rodriguez JJ, Ortega E, Garcia-Alvarez A, Brugaletta S, Sabate M, Dantas AP. Direct actions of dapagliflozin and interactions with LCZ696 and spironolactone on cardiac fibroblasts of patients with heart failure and reduced ejection fraction. ESC Heart Fail. 2023 Feb;10(1):453-464. doi: 10.1002/ehf2.14186. Epub 2022 Oct 27. PMID 36303443
- [Derived] Ortega-Paz L, Laudani C, Sionis A, Vidal-Cales P, Arevalos V, Andrea R, Morr CI, De Diego O, Ortega E, Jimenez-Trinidad FR, Dantas AP, Angiolillo DJ, Sabate M, Ortiz-Perez JT, Brugaletta S. Effect of DAPAgliflozin on Myocardial Fibrosis and Ventricular Function in Patients with ST-Segment Elevation Myocardial Infarction-DAPA-STEMI Trial. J Cardiovasc Dev Dis. 2025 Jun 11;12(6):220. doi: 10.3390/jcdd12060220. PMID 40558655